CLINICAL TRIAL: NCT00217958
Title: Better Asthma Outcomes: Lowering Tobacco Smoke Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Medical Foundation (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 295; R01HL070012 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Lung Diseases; Asthma
MeSH Terms: conditions — Lung Diseases; Asthma

INTERVENTIONS:
Behavioral: SHS reduction intervention based on social cognitive learning theory

SUMMARY:
To improve disease outcomes through reduction in secondhand tobacco smoke exposure of children with asthma

DETAILED DESCRIPTION:
BACKGROUND:

Secondhand tobacco smoke (SHS) exposure increases asthma morbidity in children. Efforts to reduce exposure have had mixed results. This study is a randomized controlled trial of an exposure reduction intervention, with objective feedback to parents on the child's exposure based on urine cotinine measurement, and counseling tailored to the child's specific exposure sources/locations and parental readiness to take specific actions to reduce exposure from each source/location. This trial involves 350 SHS-exposed children with persistent asthma, 3-12 years of age, receiving care from the Kaiser Health Care Program in Northern California. Primary outcomes over the 18 months of follow-up will be asthma acute care utilization and urine cotinine/creatine ratio. Changes in controller medication adherence will be evaluated using a pharmacy-based dispensing index.

DESIGN NARRATIVE:

Primary objective: To evaluate the efficacy of a behaviorally-based, cotinine-feedback-and-monitoring program designed to reduce SHS exposure in an 18-month randomized controlled trial (RCT) with 350 children with persistent asthma, 3-12 years of age, in comparison with usual medical care.

Secondary objectives: 1) to investigate the behavioral mechanisms that mediate between the intervention and associated improvements in asthma outcomes, and 2) to determine the influence of initial caregiver stage of change with regard to smoking practices on response to the intervention.

Hypotheses:

1. Disease outcomes: A behaviorally-based, individually-tailored intervention that emphasizes SHS exposure reduction, provides sequential feedback to the parent on the child's urine cotinine level, and is tailored to the parent's stage of change with regard to smoking practices will be associated with decreased asthma crisis care utilization and improvements in secondary disease outcomes over an 18-month follow-up period when compared with usual medical care.
2. ETS exposure: The SHS reduction intervention will be associated with lower SHS exposure at follow-up (assessed by urine cotinine/creatinine ratio), compared with usual medical care.
3. Mechanism: Decreases in urine cotinine/creatinine ratio will be instrumental in intervention-associated improvements in asthma crisis care utilization.

ELIGIBILITY:
* Age 3-12 years
* Kaiser member for >= 1 year
* >= 1 asthma care visit in prior year
* Persistent asthma likely based on prior year:

Physician diagnosis code of persistent asthma OR >= 4 beta agonist (BA) dispensing events OR >= 4 Anti-inflammatory (AI) dispensing events

* Secondhand smoke exposure by parent report.
* Parent agrees to participate in a clinical trial of a smoke exposure reduction interventio

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2002-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Wilson, Principal Investigator — Res Inst, Palo Alto Med Fdn

REFERENCES:
- [Background] Farber HJ, Wilson SR, Caine L, Bertorello L, Brown NL, Verghese S, Luna V, Quesenberry CP. Association between parent report of smoke exposure level, effect of smoke on child's asthma, and urine cotinine levels. Paper presented at the 2005 Annual Meeting of the American Thoracic Society, San Diago, CA, May 24, 2005. Proceedings of the American Thoracic Society; Vol.2 Abstracts Issue; 2005.
- [Background] Wilson SR, Brown NL, Farber HJ, Luna V, Verghese S, Caine L, Bertorello L, Quesenberry CP. Sources of and caregiver readiness to reduce secondhand smoke (SHS) exposure of children with asthma. Poster presented at the 2005 Annual Meeting of the American Thoracic Society, San Diago, CA, May 24, 2005. Proceedings of the American Thoracic Society; Vol.2 Abstracts Issue; 2005.
- [Derived] Wilson SR, Farber HJ, Knowles SB, Lavori PW. A randomized trial of parental behavioral counseling and cotinine feedback for lowering environmental tobacco smoke exposure in children with asthma: results of the LET'S Manage Asthma trial. Chest. 2011 Mar;139(3):581-590. doi: 10.1378/chest.10-0772. Epub 2010 Sep 23. PMID 20864611
- [Derived] Farber HJ, Knowles SB, Brown NL, Caine L, Luna V, Qian Y, Lavori P, Wilson SR. Secondhand tobacco smoke in children with asthma: sources of and parental perceptions about exposure in children and parental readiness to change. Chest. 2008 Jun;133(6):1367-1374. doi: 10.1378/chest.07-2369. Epub 2008 Mar 13. PMID 18339788